CLINICAL TRIAL: NCT06132919
Title: A Parallel Group (2-arm), Randomised, Double-blind, 12-week Trial to Explore the Efficacy and Safety of MC2-25 Cream and MC2-25 Vehicle in Women Diagnosed With Vulvar Lichen Sclerosus (VLS)
Brief Title: Efficacy and Safety of MC2-25 Cream & Vehicle in Women With Vulvar Lichen Sclerosus (VLS)
Acronym: Orchid 1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MC2 Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MC2-25-C3
Record Dates: First submitted 2023-11-10; First posted 2023-11-15 (Actual); Results first posted 2025-10-15 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-09

CONDITIONS: Vulvar Lichen Sclerosus
MeSH Terms: conditions — Vulvar Lichen Sclerosus

STUDY DESIGN:
Intervention Model Description: Parallel-group, Randomized, Double-blind
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MC2-25 cream (Experimental): MC2-25 cream will be applied daily for 12 weeks
  Interventions: Drug: MC2-25 cream
- MC2-25-vehicle (Experimental): MC2-25 vehicle will be applied daily for 12 weeks
  Interventions: Drug: MC2-25 vehicle

INTERVENTIONS:
Drug: MC2-25 cream — Topical application
  Arms: MC2-25 cream
Drug: MC2-25 vehicle — Topical application
  Arms: MC2-25-vehicle

SUMMARY:
The purpose of this study is to explore the efficacy and safety of MC2-25 cream and MC2-25 vehicle in women with vulvar lichen schelosus (VLS).

DETAILED DESCRIPTION:
In this study, subjects who fulfil all inclusion and exclusion criteria are enrolled.

Eligible subjects will be randomized in a 1:1 ratio to MC2-25 cream or MC2-25 vehicle, respectively.

The subjects will apply the assigned investigational medicinal product (IMP) daily for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Women, of any race or ethnicity, who are ≥18 years of age at the time of screening.
* Able to understand the trial and willing to comply with trial requirements.
* Has provided written informed consent.
* Clinical diagnosis of VLS.
* Presence of at least one of the following signs of VLS: Hyperkeratosis and/or Sclerosis.
* First symptoms of VLS noticed by the patient at least 6 months before baseline.
* At least four WI-NRS scores available in the diary for calculation of the average WI-NRS at the baseline visit.
* At least moderate itch defined as average WI-NRS ≥4 at the Baseline visit.
* Women must be of either of non-childbearing potential or childbearing potential with a negativ urine pregnancy test at baseline.
* Women of childbearing potential must agree to use a highly effective method of contraception.

Exclusion Criteria:

* Pregnant, breast feeding, or planning to become pregnant during the trial.
* Any (other than VLS) ongoing localized or systemic disease involving the vulvar region.
* Ongoing symptomatic Urinary Tract Infection.
* Ongoing or prior diagnosis of any genitoanal malignancy or pre-malignancy.
* Any kind of ongoing cancer prior to the Baseline visit.
* Any chronic or acute systemic medical condition that, in the opinion of the investigator, may pose a risk to the safety of the patient or may interfere with the assessment of efficacy in this trial.
* Known history of allergic reaction to any ingredients in MC2-25 cream or MC2-25 vehicle.
* Start of a new or change of existing non-biologic systemic treatment, within 21 days prior to the Baseline visit.
* Start of a new or change of existing biologic systemic treatment, within 3 months or 5 half-lives (whichever is longest) prior to the Baseline visit.
* Start of a new or change of existing systemic or intravaginal treatment with estrogen containing products, within 21 days prior to the Baseline visit.
* Start of new or change of menstrual care routines within 21 days prior to the Baseline visit.
* Use of emollients on the vulvar region within 3 days prior to the Baseline visit.
* Use of any topical treatment on the vulvar region, within 14 days prior to the Baseline visit.
* Use of any light therapy on the vulvar region, within 28 days prior to the Baseline visit.
* Received a non-marketed or blinded drug within 28 days or 5 half-lives (whichever is longer) prior to the Baseline visit.
* If in the opinion of the investigator, the patient is unlikely to comply with the clinical trial protocol.
* If previously randomized in this trial.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women diagnosed with vulvar lichen sclerosus (VLS) may enter the trial
Enrollment: 33 (Actual)
Dates: Start 2023-10-11 (Actual); Primary Completion 2024-11-08 (Actual); Study Completion 2024-11-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- MC2 Therapeutics study site, Kolding, Denmark

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MC2-25 Cream | MC2-25-vehicle
Started | 16 | 17
Completed | 13 | 15
Not Completed | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MC2-25 Cream | MC2-25-vehicle | Total
Number analyzed (Participants) | 16 | 17 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.1 (14.3) | 57.5 (14.5) | 54.9 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 17 | 33
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 15 | 17 | 32
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 15 | 17 | 32
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Denmark | 16 | 17 | 33

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Weekly Mean Worst Itch Numeric Rating Score (WI-NRS)
Description: Mean change in weekly Worst Itch Numeric Rating score WI-NRS (as measured on a 11-point numeric rating scale from 0 - 10, where 0 represents no itch and 10 represents worst imaginal itch), calculated as the average of weekly means WI-NRS values from Baseline to Week 12 for MC2-25 cream compared to MC2-25 vehicle.
Time Frame: 12 weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | MC2-25 Cream | MC2-25-vehicle
Number analyzed (Participants) | 16 | 17
units on a scale | -4.0 (0.8) | -3.5 (0.7)

ADVERSE EVENTS:
Time Frame: Adverse event information was collected from individual trial subjects from signature of the informed consent form and until the last trial visit, up to 18 weeks.
Description: Out of the 33 randomized subjects, 1 subject did not receive any treatment. The overall number of treated subjects, and thus included in the Adverse Event summary is 32 subjects (15 in the MC2-25 Cream group and 17 in the MC2-25-vehicle group.
Arm/Group | MC2-25 Cream | MC2-25-vehicle
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/17
Other Adverse Events (participants affected / at risk) | 11/15 | 15/17
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MC2-25 Cream (N=15) | MC2-25-vehicle (N=17)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anal fissure (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Application site disconfort (General disorders) | 1 (1) | 0 (0)
Application site pain (General disorders) | 4 (6) | 6 (7)
Application site pruritus (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Acarodermatitis (Infections and infestations) | 0 (0) | 1 (1)
Anal fungal infection (Infections and infestations) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 2 (2)
Eye infection (Infections and infestations) | 0 (0) | 1 (1)
Herpes simplex (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 3 (3) | 3 (3)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1)
Pelvic inflammatory disease (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2) | 1 (1)
Tinea infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 3 (6) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vulvovaginal injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vitamin D decreased (Investigations) | 1 (1) | 0 (0)
Calcium deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1) | 1 (1)
Incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Genital haemorrhage (Reproductive system and breast disorders) | 1 (1) | 2 (2)
Lichen Sclerosis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Menstrual disorder (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vulval oedema (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vulvovaginal burning sensation (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vulvovaginal erythema (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vulvovaginal pain (Reproductive system and breast disorders) | 4 (4) | 2 (3)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 3 (3) | 2 (2)
Vulvovaginal rash (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Nail disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3)
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2024-07-31): https://cdn.clinicaltrials.gov/large-docs/19/NCT06132919/Prot_000.pdf
  • Statistical Analysis Plan (2024-10-30): https://cdn.clinicaltrials.gov/large-docs/19/NCT06132919/SAP_001.pdf